CLINICAL TRIAL: NCT05178017
Title: Effectiveness of the Lifestyle Eating and Performance (LEAP) Program for the Treatment of Irritable Bowel Syndrome (IBS)
Brief Title: Lifestyle Eating and Performance (LEAP) Program for the Treatment of Irritable Bowel Syndrome (IBS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Biomedical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00048988
Record Dates: First submitted 2021-10-25; First posted 2022-01-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants (Experimental): Individuals with Irritable Bowel Syndrome (IBS)
  Interventions: Diagnostic Test: Leukocyte Activation Assay (LAA-MRT) / Lifestyle Eating and Performance (LEAP) program

INTERVENTIONS:
Diagnostic Test: Leukocyte Activation Assay (LAA-MRT) / Lifestyle Eating and Performance (LEAP) program — The LEAP program is based on the in-vitro Leukocyte Activation Assay (LAA-MRT) results and initially prepared with the least immune reactive foods and chemicals, and subsequent foods will be added depending on the degree of immune reactivity in a nutritionally balanced manner.

SUMMARY:
A three month follow-up study to evaluate the effectiveness of a tailored anti-inflammatory eating plan guided by a registered dietitian to treat irritable bowel syndrome.

DETAILED DESCRIPTION:
This study will have 60 participants with Irritable bowel syndrome (IBS) for a duration of three months. The procedures will consist of anthropometric measures, blood pressure, questionnaires, and a blood sample. There will be seven visits with one including a virtual meeting with a registered dietitian involved in the Lifestyle Eating and Performance (LEAP) program. With these procedures the investigators will test the effectiveness of the LEAP program for the treatment of irritable bowel syndrome by improving inflammatory markers, symptoms, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an established diagnosis of IBS-D as determined by Rome III or IV Criteria
* Have IBS of at least moderate severity
* Must be on a stable dose regimen for at least 1 month prior to enrollment
* Willing to follow the LEAP program for 3 months
* Able to give informed consent
* Willing to complete the study

Exclusion Criteria:

* Individuals with a history of inflammatory bowel disease, celiac disease, abdominal surgeries, cancer patients under treatment, and kidney failure
* BMI of 40 or higher
* Pregnancy or planned pregnancy or lactation
* Any serious illness that will interfere with the study procedures or results
* Enrollment in active clinical trial/ experimental therapy within the last 30 days
* Currently on another dietary treatment approach

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory blood markers | 3 months
  To evaluate the cytokines levels (IL-I b; IL-6; IL-8; IL-10; IL-12; IL-17; TNF-a) of participants with irritable bowel syndrome from baseline levels to 12 weeks by using a Bio-Plex 200 System (Bio-Rad, California, USA).

SECONDARY OUTCOMES:
Gastrointestinal symptoms severity | 3 months
  To evaluate gastrointestinal symptoms severity of participants with irritable bowel syndrome from baseline to 12 weeks by using the IBS-Symptom Severity Scale (IBS-SSS). Items relate to gastrointestinal pain, bowel dysfunction, and overall wellbeing will be used to evaluate IBS severity. A higher score indicating worse condition.
The quality of life | 3 months
  To evaluate the quality of life of participants with irritable bowel syndrome from baseline to 12 weeks using the IBS-36 Quality of Life (IBS-36): The self-administrated IBS-36 questionnaire consists of 36 individual questions. Each question's response is scored on a 7-point Likert scale where 0 = never and 6 = always. A final score is a sum of the scores of the 36 questions. The highest possible score on the IBS-36 is 216, and the lowest is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Zarini, Ph.D., RD, Principal Investigator — Oxford Biomedical Technologies, Inc.
Locations (1):
- Oxford Biomedical Technologies, Inc., Riviera Beach, Florida, United States